CLINICAL TRIAL: NCT00129337
Title: A Multicenter, Open-Label Safety and Pharmacokinetics Study of Chimeric Anti-Phosphatidylserine Monoclonal Antibody (Bavituximab) in Patients With Refractory Advanced Solid Tumor Malignancies
Brief Title: Study of Bavituximab in Patients With Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Jennifer Lai, MBA, CCRA, Peregrine Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0401
Expanded Access: Available
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Tumors
Keywords: monoclonal antibody; phase 1; solid tumor; anti-angiogenesis; refractory advanced solid tumor malignancy
MeSH Terms: conditions — Neoplasms | interventions — bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 0.1 mg/kg
  Interventions: Drug: Bavituximab
- 2 (Experimental): 0.3 mg/kg
  Interventions: Drug: Bavituximab
- 3 (Experimental): 1 mg/kg
  Interventions: Drug: Bavituximab
- 4 (Experimental): 3 mg/kg
  Interventions: Drug: Bavituximab

INTERVENTIONS:
Drug: Bavituximab — Bavituximab is a sterile drug solution supplied in glass bottles. Bavituximab will be intravenously administered over approximately 90 minutes on days 0, 7, 14 and 21 (dosage determined based on dose cohort and body weight).

SUMMARY:
The purpose of this study is to determine the safety of bavituximab when administered via a vein, and to examine how bavituximab behaves in the body - how quickly it is taken up by the body and how long it stays there. The effect of bavituximab on tumor responses will also be examined.

DETAILED DESCRIPTION:
The genetic variations observed in most advanced cancers decrease the effectiveness of many anti-cancer agents through the development of drug resistance. Therefore, alternative approaches to the direct targeting of cancer cells are urgently needed. Bavituximab is the generic name for a chimeric (human/murine) monoclonal antibody directed against aminophospholipids. Bavituximab is Peregrine's first investigational product under its anti-phospholipid therapy technology platform. Anti-phospholipid therapy is a novel approach to treating cancer. It is based on the finding that aminophospholipids, which are basic components of the inner surface of cells become externally exposed in response to certain disease states such as cancer. Laboratory and animal studies have demonstrated that bavituximab specifically targets cancer cells and inhibits tumor growth in a variety of experimental cancer models. This study will examine the safety and tolerability of bavituximab when administered to patients with advanced solid tumor cancers that are unresponsive to current therapies. Cohorts of 6 patients each will be treated at the starting dose of 0.1 mg bavituximab per kilogram body weight (0.1 mg/kg). Successive patient cohorts will receive 0.3, 1.0 and 3.0 mg/kg of bavituximab. Patients will be followed for a total of 56 days. Patients who demonstrate an objective tumor response will be offered further bavituximab treatment on an extension protocol.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age with life expectancy of 3 months
* Evaluable, histologically or cytologically confirmed, refractory advanced solid tumor malignancy
* ECOG score of less than or equal to 1
* Adequate hematologic function (absolute neutrophil count [ANC] greater than or equal to 1,500 cells/uL; hemoglobin greater than or equal to 9 g/dL; platelets greater than or equal to 100,000/uL and less than or equal to 500,000/uL)
* Adequate renal function (serum creatinine less than or equal to 1.5 mg/dL or calculated creatinine clearance greater than 60 mL/min)
* Adequate hepatic function (bilirubin less than or equal to 1.5 x ULN; ALT less than or equal to 3 x ULN; AST less than or equal to 3 x ULN)
* Normal coagulation profile (prothrombin time/international normalized ratio [PT/INR] and activated partial thromboplastin time [aPTT] within institutional normal limits)
* D-dimer less than or equal to 2 times upper limit of institutional normal
* New York Heart Association classification I or II for patients with significant cardiopulmonary disease
* Female patients must have a negative serum pregnancy test at prestudy and all patients of reproductive potential must be willing to use an approved form of barrier method contraception

Exclusion Criteria:

* Prior exposure to any chimeric antibody
* Any evidence of clinically significant bleeding
* Known history of bleeding diathesis or coagulopathy
* Any history of thromboembolic events including central venous catheter-related thrombosis within the past 12 months
* Any evidence or history of hypercoagulable state (eg, shortened aPTT)
* Concurrent therapy with oral or parenteral anticoagulants
* Concurrent hormone therapy (ie, estrogen contraceptives, hormone replacement, anti-estrogen)
* Chemotherapy, immunotherapy or radiotherapy within 4 weeks of day 0 (6 weeks for nitrosoureas and mitomycin C) or have not recovered from treatment-related side effects due to agents administered more than 4 weeks earlier (stable, non-hematological residual toxicities of Grade 1 or less and Grade 2 dry skin or alopecia are allowed)
* Investigational therapy within 4 weeks of day 0
* Evidence of central nervous system (CNS) metastatic disease at prestudy (no active brain metastases on magnetic resonance imaging [MRI] at prestudy)
* Major surgery within 4 weeks of day 0
* Pregnant or nursing women
* Uncontrolled intercurrent disease (eg, diabetes, hypertension, thyroid disease)
* Any history of angina pectoris, coronary artery disease or cerebrovascular accident, or transient ischemic attack
* A history of any condition requiring anti-platelet therapy with the exception of general cardiovascular prophylaxis with aspirin
* A history of any condition requiring treatment (past or current) with coumarin-type agents within the past 12 months
* Cardiac arrhythmia requiring medical therapy
* Serious non-healing wound
* Requirement for chronic daily treatment with non-steroidal anti-inflammatory drugs (NSAIDs), anti-platelet drugs (eg, phosphodiesterase inhibitors, adenosine diphosphate receptor antagonists) or steroids
* Known chronic infection with HIV or hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
adverse events | Study Completion
laboratory evaluations | Study Completion
human anti-chimeric antibody | Study Completion
pharmacokinetic analysis | Study Completion

SECONDARY OUTCOMES:
tumor evaluation by Response Evaluation Criteria in Solid Tumors (RECIST) | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Nuhad Ibrahim, MD, Principal Investigator — M.D. Anderson Cancer Center; Linda Garland, MD, Principal Investigator — University of Arizona; Lee Rosen, MD, Principal Investigator — Premiere Oncology, A Medical Corporation (Santa Monica); Lucas Wong, MD, Principal Investigator — Scott & White Memorial Hospital; Lee S Schwartzberg, MD, FACP, Principal Investigator — The West Clinic; David E Gerber, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (6):
- United States (6):
  - Arizona Cancer Center, Tucson, Arizona
  - Premiere Oncology, Santa Monica, California
  - The West Clinic, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Scott & White Hospital, Center for Cancer Prevention and Care, Temple, Texas